CLINICAL TRIAL: NCT07295236
Title: Prospective Observational Study on Endo-vac Therapy for Esophago-jejunal Anastomotic Leak
Brief Title: Impact of Endo-vac Therapy for Esophago-jejunal Anastomotic Leak
Acronym: ENDO-VAL
Status: Recruiting | Type: Observational
Sponsor: Ukrainian Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Oleksii Dobrzhanskiy, Surgical oncoligist, Ukrainian Society of Clinical Oncology
Other Study IDs: 9947/2025
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Esophagojejunal Anastomotic Leak
Keywords: gastric cancer; esophagojejunal anastomotic leak; total gastrectomy; Endoscopic vacuum therapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endo-vac cohort: Patients who are diagnosed with asophago-jejunal anastomotic leakage will undergo endoscopic vacuum therapy. Local source control may be additionally achieved with para-anastomotic drains.

SUMMARY:
The goal of this observational study is to assess the impact of endoscopic vacuum therapy in patients who underwent total gastrectomy due to gastric cancer and developed esophago-jejunal anastomotic leakage. The main outcomes to be investigated are the following:

Primary endpoint: mortality rate Secondary endpoints: morbidity rate, time from AL diagnosis to discharge, patients satisfactory rate.

DETAILED DESCRIPTION:
Patients who are diagnosed with asophago-jejunal anastomotic leakage will undergo endoscopic vacuum therapy. Local source control may be additionally achieved with para-anastomotic drains.

ELIGIBILITY:
Inclusion Criteria:

* patients who developed esophago-jejunal anastomotic leak less than 50% of circumference of anastomosis
* patients who developed esophago-jejunal anastomotic leak and remained stable at the moment of diagnosis with no indications for diversion surgery

Exclusion Criteria:

* unstable patients who developed esophago-jejunal anastomotic leak
* patients who developed esophago-jejunal anastomotic leak more than 50% or anastomotic circumference
* patients who rejected endoscopic vacuum therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population involves ukrainian patients who developed esophago-jejunal anastomotic leak after total gastrectomy due to gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 90 days after last endo-vac placement
  Mortality rate associated with endoscopic vacuum therapy

SECONDARY OUTCOMES:
Morbidity rate | 90 days after last endoscopic vacuum placement
  Rate of complications associated with endoscopic vacuum therapy or ineffective local control
Time from AL diagnosis to discharge | The number of days from from AL diagnosis to discharge
  time from AL diagnosis to discharge
Patients satisfactory rate | 90 days after discharge, 365 days after discharge, 2/3/4/5 years after discharge
  Patients satisfactory rate assessed by quality of life questionnaires and patient-reported outcomes scales

CONTACTS AND LOCATIONS:
Overall Officials: Oleksii Dobrzhanskyi, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Anonymous IPD will be shared upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code